CLINICAL TRIAL: NCT07254598
Title: Efficacy of Myotensive Techniques Applied to the Extraocular Muscles as an Adjunct to Manual Therapy in the Treatment of Migraine Without Aura
Brief Title: Myotensive Extraocular Muscle Techniques Added to Manual Therapy for Migraine Without Aura
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Facultad de Enfermería, Fisioterapia y Podología (FEFP) (Other)
Responsible Party: Principal Investigator, Dr. María de la Casa Almeida, PhD, Physiotherapist, University of Seville., Facultad de Enfermería, Fisioterapia y Podología (FEFP)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECAOJO
Record Dates: First submitted 2025-11-13; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Migraine Without Aura
Keywords: migraine; Oculomotor Muscles; Musculoskeletal Manipulations; Physical Therapy Services
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is considered double-blind because two levels of blinding are implemented:
  Blinding of participants:
  Subjects will not know whether they are receiving the experimental intervention (cranio-cervical manual therapy combined with extraocular myotensive techniques) or the control intervention (standard cranio-cervical manual therapy only). To achieve this, both interventions will be applied under identical conditions of duration, frequency, environment, and therapist-patient contact, so that the subjective treatment experience remains indistinguishable and participants cannot identify which group they belong to.
  Blinding of outcome assessors:
  The physiotherapists and optometrists responsible for performing pre- and post-intervention measurements will not know the participants' group allocation. Data will be coded and analyzed using numerical identifiers to ensure objectivity in the evaluation of results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myotensive Extraocular Muscle Techniques + Manual Therapy (Experimental): Cranio-Cervical Manual Therapy Combined with Extraocular Myotensive Techniques
  Interventions: Other: Myotensive Extraocular Muscle Techniques + Manual Therapy
- Standard Manual Therapy (Active Comparator): Standard Cranio-Cervical Manual Therapy
  Interventions: Other: Standard Manual Therapy

INTERVENTIONS:
Other: Myotensive Extraocular Muscle Techniques + Manual Therapy — This intervention consists of six 55-minute sessions over eight weeks. It combines standard cranio-cervical manual therapy techniques-such as suboccipital inhibition, cervical traction, vertebral segmental mobilization, and temporomandibular joint decompression-with specific myotensive techniques applied to the extraocular muscles. The oculomotor component is performed in a supine position, using gentle isometric and eccentric tension-release maneuvers targeted to the most restricted eye movement directions. The goal is to modulate extraocular muscle tone, optimize the cervico-ocular proprioceptive relationship, and reduce migraine-related dysfunctions.
  Arms: Myotensive Extraocular Muscle Techniques + Manual Therapy
Other: Standard Manual Therapy — This intervention consists of six 40-minute sessions over eight weeks, matching the experimental group in duration, frequency, and clinical environment. It includes suboccipital inhibition, cervical traction, segmental vertebral mobilization, and temporomandibular joint decompression techniques. No ocular or visual system intervention is performed. The purpose is to serve as an active control for the cranio-cervical component of the treatment.
  Arms: Standard Manual Therapy

SUMMARY:
Migraine without aura is a highly prevalent and disabling primary headache that significantly affects quality of life. Many patients experience insufficient symptom control with pharmacological treatments or develop adverse effects, which has increased interest in safe, non-invasive therapeutic alternatives. Physiotherapy, and particularly manual therapy, has shown potential benefits in reducing pain and improving function in headache disorders. This randomized clinical trial will evaluate the effectiveness of adding specific myotensive techniques directed at the extraocular muscles to a craniocervical manual therapy program in adults with migraine without aura. The hypothesis is that targeting the oculomotor system may influence pain modulation and improve symptoms related to visual, cervical, and sensorimotor interactions.

Ninety participants aged 18 to 65 years with a medical diagnosis of migraine without aura according to the International Classification of Headache Disorders, Third Edition (ICHD-III), will be randomly assigned to an experimental group or a control group. Both groups will receive six physiotherapy sessions over approximately eight weeks. The experimental group will receive manual therapy on the craniocervical region and temporomandibular joint (TMJ) combined with myotensive techniques for the extraocular muscles, while the control group will receive only the standard manual therapy protocol. Evaluations will be conducted at baseline and post-intervention using validated instruments such as the Migraine Disability Assessment (MIDAS), Craniofacial Pain and Disability Inventory (CF-PDI), Migraine-Specific Quality of Life Questionnaire (MSQ), and Visual Analogue Scale (VAS) for pain. Cervical mobility and oculomotor function will also be assessed through standardized clinical tests.

All procedures will be carried out at the Faculty of Nursing, Physiotherapy and Podiatry of the University of Seville. Data will be collected and managed in digital format in compliance with the General Data Protection Regulation (GDPR) and Spanish data protection law. Study results are expected to clarify the role of the oculomotor system in migraine without aura and to determine whether incorporating extraocular myotensive techniques enhances the effects of manual therapy within a comprehensive physiotherapeutic approach.

DETAILED DESCRIPTION:
Migraine without aura is a complex neurological condition involving interactions between sensory, musculoskeletal, and central regulatory systems. Its recurrent pain episodes, associated symptoms, and functional impact make it a major cause of disability. Despite therapeutic advances, a substantial proportion of patients continue to experience insufficient symptom control or intolerance to medication, reinforcing the need for complementary, non-pharmacological treatment strategies. Physiotherapy, and specifically manual therapy, has gained increased relevance due to its safety, individualized application, and potential influence on neuromuscular and sensorimotor mechanisms involved in migraine.

Alterations in the craniocervical region, including muscular hypertonicity, reduced mobility, and altered proprioception, are frequently observed in patients with migraine. These factors may contribute to pain modulation and central sensitization. Within this context, the oculomotor system has emerged as an area of interest due to its strong anatomical and functional connections with the upper cervical spine, brainstem integration centers, and vestibular and proprioceptive pathways. Extraocular muscles provide continuous proprioceptive input essential for coordinating gaze and head orientation. Dysfunction in this system may affect sensory integration, postural control, and cervico-ocular interactions, potentially contributing to increased sensory load and symptom exacerbation.

Myotensive techniques applied to the extraocular muscles aim to regulate muscle tone, optimize ocular motility, and influence afferent sensory input to central integration centers. When combined with manual therapy directed at the craniocervical region and temporomandibular joint (TMJ), these techniques may contribute to improving neuromuscular coordination and reducing migraine-related symptoms. This trial seeks to evaluate the clinical effects of incorporating extraocular myotensive techniques into a structured manual therapy program in patients with migraine without aura.

The study is a randomized, controlled, parallel-group clinical trial designed to compare two physiotherapy interventions. Ninety participants aged 18 to 65 years with a medical diagnosis of migraine without aura according to the International Classification of Headache Disorders, Third Edition (ICHD-III), will be randomly assigned through a computer-generated sequence to an experimental group or a control group. An independent researcher will manage allocation concealment using opaque, sealed envelopes. Evaluators will be blinded to group assignment, and data analysis will be conducted under blinded conditions.

Both groups will receive six physiotherapy sessions over approximately eight weeks. The experimental group will receive combined craniocervical manual therapy and specific myotensive techniques applied to the extraocular muscles. The control group will receive the same craniocervical manual therapy program without oculomotor techniques. All interventions will be administered by physiotherapists trained in manual therapy. Oculomotor assessments will be supervised by professionals with expertise in optometry.

Outcome measures will be assessed at baseline and post-intervention. Pain and disability will be evaluated through validated instruments, including the Visual Analogue Scale (VAS), Migraine Disability Assessment (MIDAS), Craniofacial Pain and Disability Inventory (CF-PDI), and the Migraine-Specific Quality of Life Questionnaire (MSQ). Cervical range of motion will be assessed using a gravity goniometer. Neuromuscular function of the deep cervical flexors will be evaluated through the Cranio-Cervical Flexion Test (CCFT) using pressure biofeedback in millimeters of mercury (mmHg), generating the Activation Score (AS) and Performance Index (PI). Oculomotor evaluation will include assessment of ocular motility, gaze-related pain perception, and functional changes in different gaze directions. Postural alignment of the head will be measured using goniometric procedures in a relaxed standing position. Heterophoria will be quantified using the Von Graefe test, expressed in prism diopters (Δ), with results categorized into esophoria (base-out, BO) or exophoria (base-in, BI) as applicable.

All study procedures will take place at the Faculty of Nursing, Physiotherapy and Podiatry of the University of Seville. Data collection will be performed exclusively through secure digital platforms, ensuring compliance with the General Data Protection Regulation (GDPR) and relevant Spanish legislation on personal data protection. The intervention is non-pharmacological and low-risk, and all participants will provide written informed consent prior to enrollment.

The purpose of this clinical trial is to determine whether incorporating specific techniques directed at the extraocular muscles enhances the effects of manual therapy in patients with migraine without aura. By examining changes in pain intensity, migraine frequency, disability, quality of life, cervical function, and oculomotor performance, this study aims to contribute new evidence to physiotherapy-based approaches and expand the range of safe and effective therapeutic options for individuals living with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Being of legal age.
* Having a medical diagnosis of migraine without aura established by a neurologist, according to the criteria of the ICHD-III
* Having been diagnosed with migraine for at least one year and experiencing at least one attack per month.
* Having been prescribed a specific pharmacological treatment by a specialist physician for at least 6 months.
* Participants must attend all assessments with their habitual optical correction fully updated (glasses or contact lenses), ensuring that any refractive error is appropriately corrected.
* Presenting symptoms in the oculomotor system, as detailed in the participant information sheet.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Receiving any other type of physiotherapeutic treatment at the time of the intervention.
* Presenting any of the following conditions: chronic respiratory, cardiovascular, and/or musculoskeletal diseases such as polyarthritis, rheumatic muscle inflammation, osteoporosis, or osteoarthritis; other types of headache, other neurological diseases, oncological processes, cognitive, emotional, or psychological disorders; previous surgical interventions or trauma in the cervical region; or diseases specific to the oculomotor system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline (pre-intervention, prior to the first treatment session) and immediately after each treatment session, through study completion.
  This continuous quantitative variable assesses the intensity of pain experienced by the patient. The VAS consists of a 10 cm horizontal line whose endpoints are anchored by the expressions "no pain" on the left end and "worst pain imaginable" on the right end. The patient is asked to mark the point along this line that best represents their subjective perception of pain at that moment, and the score is obtained by measuring in centimeters from the left end to the mark made.
Score obtained from the Craniofacial Pain and Disability Inventory (CF-PDI) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  This discrete quantitative variable, originally named the Craniofacial Pain and Disability Inventory (CF-PDI), is a questionnaire specifically designed to assess pain and disability in patients suffering from craniofacial pain, such as headaches, temporomandibular disorders, and related conditions.
  The aim of the questionnaire is to evaluate the severity of craniofacial pain and its impact on patients' functional, emotional, and social activities.
  It is structured into items grouped into four dimensions: the impact on daily activities, work, interpersonal relationships, and emotional state. Each item is rated on a 5-point Likert scale ranging from 0 to 4, where 0 indicates minimal impact and 4 indicates maximum perceived impact in each dimension. The total score can reach up to 84 points, with higher scores reflecting greater levels of disability and impact of craniofacial pain on the patient's life.
  This tool has demonstrated excellent psychometric properties, with high reliability i
Score obtained from the Migraine-Specific Quality of Life Questionnaire (MSQ) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  This continuous quantitative variable corresponds to a tool used to assess the impact of migraine on patients' quality of life. The MSQ includes 14 items that explore the frequency and intensity of migraine episodes and their impact on work activities, social relationships, emotional well-being, and overall health status. Responses are rated using a Likert-type scale.
  The questionnaire is divided into subscales corresponding to different domains of life affected by migraine: physical functioning, emotional functioning, and social functioning. The total score is obtained by summing the subscale scores.
  Each of the 14 items is rated on a 6-point Likert scale ranging from 1 = "all the time" to 6 = "never," thus evaluating how frequently migraine interferes with different aspects of the patient's life.
  To facilitate interpretation and standardization, raw scores from the MSQ are transformed to a standardized 0-100 scale. This transformation is achieved by subtracting the minimum possible
Score obtained from the Short Form-36 Health Survey (SF-36) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  This continuous quantitative variable is used to measure health-related quality of life, encompassing multiple aspects of physical and mental well-being. The SF-36 consists of 36 items divided into eight subscales evaluating different dimensions of health: Physical Functioning (PF), Social Functioning (SF), Role Emotional (RE), Vitality (VT), Mental Health (MH), Bodily Pain (BP), General Health (GH), and Physical Health (PH). Each subscale is scored from 0 to 100, where higher scores indicate better quality of life in that particular domain. Subscale scores can be analyzed individually or combined to generate an overall quality of life index.
  The SF-36 was developed by Ware et al. (1992) and adapted and validated into Spanish as part of the international IQOLA project by Vilagut et al. The SF-36 has demonstrated excellent reliability and validity across diverse populations and clinical contexts. It shows high internal consistency, with Cronbach's alpha coefficients generally above 0.8
Score obtained from the Migraine Disability Assessment Questionnaire (MIDAS) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  This continuous quantitative variable is a self-administered tool designed to evaluate the impact of migraine on patients' daily activities over the past three months. It consists of five questions assessing the number of days lost in work, household, and social activities due to migraine. The total score is obtained by summing responses to these five questions and is classified into four disability grades: 0-5 points: little or no disability 6-10 points: mild disability 11-20 points: moderate disability ≥21 points: severe disability Additionally, the questionnaire includes two supplemental questions that gather information on the frequency of migraine episodes and the average pain intensity on a 0-10 scale. The MIDAS has shown moderately high test-retest reliability and good convergent validity.
Score obtained from the Headache Impact Test (HIT-6) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  This continuous quantitative variable consists of a questionnaire with six items assessing the impact of headaches across various aspects of a patient's life, including pain, functional limitation, fatigue, cognition, and emotional status, providing a global overview of headache burden. Each item is rated on a 5-point frequency scale: never (6 points), rarely (8 points), sometimes (10 points), very often (11 points), and always (13 points).
  The total score ranges from 36 to 78 and is interpreted as follows:
  ≤49: little or no impact 50-55: some impact 56-59: substantial impact
  ≥60: severe impact The HIT-6 has demonstrated excellent psychometric properties, with internal consistency (Cronbach's alpha) ranging from 0.78 to 0.90 across studies, strong validity through correlations with other migraine assessment scales such as MIDAS and SF-36, and high reproducibility, with test-retest coefficients above 0.80.

SECONDARY OUTCOMES:
Cervical Range of Motion - Flexion and Extension | before first session and immediately after each of the 6 treatment sessions
  This continuous quantitative variable will be measured using a gravity goniometer, expressed in degrees. Participants will be asked to actively perform flexion and extension movements. Three measurements will be taken, and the mean value will be recorded.
  The gravity goniometer has demonstrated validity and reliability for assessing cervical range of motion, with excellent intra-rater reliability (ICC > 0.85) according to Youdas et al., and good concurrent validity when compared to three-dimensional systems (differences < 5°). It also shows adequate inter-rater reliability when standardized protocols are followed.
Cervical Range of Motion - Right and Left Lateral Flexion | before first session and immediately after each of the 6 treatment sessions
  This continuous quantitative variable will be measured in degrees using a gravity goniometer. Participants will be asked to actively perform right (RSB) and left (LSB) lateral flexion movements three times each, and the mean value will be calculated.
Cervical Range of Motion - Right and Left Rotation | before first session and immediately after each of the 6 treatment sessions
  This continuous quantitative variable will be measured in degrees using a gravity goniometer. Participants will be asked to actively perform right (RR) and left (LR) cervical rotation three times each, and the mean value will be obtained
Cranio-Cervical Flexion Test - Activation Score (AS) | before first session and immediately after each of the 6 treatment sessions
  Assessed using the Cranio-Cervical Flexion Test (CCFT) with the Chattanooga Stabilizer™ pressure biofeedback device. The Activation Score reflects the highest pressure level (in mmHg) that the participant can achieve and maintain with correct deep cervical flexor activation and without recruitment of superficial musculature.
Cranio-Cervical Flexion Test - Performance Index (PI) | Baseline (before first session) and immediately after each of the 6 treatment sessions.
  Assessed using the Cranio-Cervical Flexion Test (CCFT) with the Chattanooga Stabilizer™ pressure biofeedback device. The Performance Index represents the product of the pressure level achieved and the duration maintained, providing a quantitative measure of deep cervical flexor endurance and control.
Head Postural Deviation in Neutral Standing Position | before first session and immediately after each of the 6 treatment sessions
  This categorical quantitative variable measures the spontaneous tilt or rotation of the head axis relative to the vertical plane in relaxed standing posture, while the participant fixates on a target 50 cm away at eye level.
  Measured with a gravity goniometer and categorized as:
  * Category 0: symmetrical position (0°)
  * Category 1: mild deviation (1°-4°)
  * Category 2: moderate deviation (5°-9°)
  * Category 3: severe deviation (≥10°)
Pain Sensation in Each Gaze Position | before first session and immediately after each of the 6 treatment sessions
  This dichotomous qualitative variable records the presence or absence of pain during eye movement or fixation in each of the nine gaze positions: primary gaze, dextroversion, levoversion, supraversion, infraversion, dextroelevation, levoelevation, dextrodepression, and levodepression.
  The examiner asks the participant to look at a target placed in each position for 4 seconds, noting any painful sensation. This helps detect patterns of oculomotor dysfunction and serves as an indirect clinical indicator of tension or hypertonicity in extraocular muscles
Ocular Motility Assessment | Before first session and immediately after each of the 6 treatment sessions
  This ordinal qualitative variable assesses whether the participant can perform complete and unrestricted eye movements in all nine gaze directions.
  The evaluation follows a standardized clinical observation using the "H-test" or star pattern, with a pen, pointer, or finger moved at approximately 50 cm distance.
  Each gaze direction is categorized as:
  * 0: full and symmetrical movement without restrictions or compensatory saccades
  * 1: incomplete movement or mild hypofunction, requiring saccades to reach the target
  * 2: clearly limited or absent movement
Modulation of Ocular Motility After Head Postural Correction in Standing Position | Before first session and immediately after each of the 6 treatment sessions
  This dichotomous ordinal qualitative variable records whether there is a symptomatic improvement (pain reduction and/or increased ocular mobility) after manual correction of head posture in neutral standing.
  Categorized as:
  * 0: no change in symptoms or ocular motility
  * 1: improvement in symptoms and/or ocular motility range
Thorington test for Heterophoria | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  The Thorington test will be used to measure latent ocular deviation, expressed in prism diopters (∆), through optical dissociation with a Maddox rod and direct reading on a calibrated scale. This method provides high intra-examiner, inter-examiner, and test-retest reliability, and is sensitive to small changes following an intervention. Its internal validity relies on strict standardization of distance, illumination, rod orientation, and accommodative demand, while its external validity is supported by its widespread use as a reference test in binocular vision research. Due to its consistency, reproducibility, and clinical relevance, the Thorington test is considered an appropriate and reliable variable for use in a clinical trial.
Alternate Cover Test with Prism Bar for Oculomotor Deviation | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  This continuous quantitative variable quantifies heterophoria in prism diopters (Δ), positive for exophoria and negative for esophoria, by neutralizing ocular recovery movement with increasing prism strength.
  Normal values: ≤4Δ at distance and ≤6Δ at near (horizontal); ≤1Δ (vertical). Reliability: moderate to high (ICC 0.65-0.90), good concurrent validity with the Von Graefe test.
Fusional Vergence Amplitude (Positive and Negative) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  Continuous quantitative variable that measures the ability of the visual system to maintain binocular fusion in response to retinal disparity stimuli induced by prisms.
  * Positive fusional vergence (convergence): base-out (BO) prisms.
  * Negative fusional vergence (divergence): base-in (BI) prisms. Values are expressed in prism diopters (Δ), recording break and recovery points.
  Normal ranges:
  * Distance: convergence ≥15Δ break / ≥10Δ recovery; divergence ≥5Δ / ≥3Δ.
  * Near: convergence ≥20Δ / ≥15Δ; divergence ≥12Δ / ≥7Δ. Test-retest reliability: ICC > 0.80.
Vertical Fusional Vergence (VV) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  Continuous quantitative variable representing the visual system's ability to maintain vertical alignment under dissociative stimuli using base-up (BU) and base-down (BD) prisms.
  Normal values: break 2-3Δ, recovery ≥1.5Δ, symmetrical between eyes. Test-retest reliability: high, with strong clinical validity.
Vergence Facility (VF) | Baseline (pre-intervention, prior to the first treatment session) and immediately after completion of the final treatment session.
  Continuous quantitative variable evaluating the efficiency of alternating between convergence and divergence. Measured in cycles per minute (cpm) using a prism combination of 3Δ base-in (BI) and 12Δ base-out (BO).
  Normal values: ≥12 cpm (near vision), ≥10 cpm (distance). Test-retest reliability: ICC > 0.75; sensitive to improvements after visual therapy.

OTHER OUTCOMES:
Participant's Sex | Baseline (at enrollment, prior to any intervention)
  This qualitative nominal variable records the sex of each participant as registered in the electronic clinical history.
Participant's Age | Baseline (at enrollment, prior to any intervention).
  This continuous quantitative variable records age in full years, calculated from the participant's date of birth. If required for specific statistical analyses, this variable may be categorized into age ranges to explore possible differences in migraine frequency, intensity, or characteristics across age groups
History of Migraine | Baseline (at enrollment, prior to any intervention).
  This nominal qualitative variable indicates whether a family history of migraine is present (Yes/No). For positive cases, the degree of kinship of the affected relative will be specified.
Medication use | Daily throughout the 8-week intervention period
  This nominal qualitative variable records the type of medication taken to reduce migraine symptoms, categorized as follows:
  * Analgesic (e.g., paracetamol/acetaminophen)
  * Specific anti-migraine medication (triptans)
  * Non-steroidal anti-inflammatory drugs (NSAIDs)
  * Antiemetic
  * Other medications
Amount of Medication Consumed | Daily throughout the 8-week intervention period
  This continuous quantitative variable records the quantity of medication consumed during a migraine attack, expressed in milligrams (mg) or number of doses per day.
Migraine Attack Intensity | Daily throughout the 8-week intervention period
  This ordinal quantitative variable records the subjective intensity of each migraine attack using a 10-point numeric rating scale, where 1 = minimal pain and 10 = maximum pain experienced.
Presence of Prodrome Prior to the Attack | Daily throughout the 8-week intervention period
  This dichotomous qualitative variable records the presence (Yes/No) of prodromal symptoms prior to the onset of a migraine episode, as well as their type when present.
Dietary Factors | Daily throughout the 8-week intervention period
  This dichotomous nominal qualitative variable records whether the participant consumed any of the following potential dietary triggers within the 24 hours prior to symptom onset: chocolate, dairy products, monosodium glutamate, caffeine, and/or histamine-rich foods.
  Participants receive an informational sheet (Annex 2) describing which foods to avoid or monitor.
Water Intake | Daily throughout the 8-week intervention period
  This continuous quantitative variable records the approximate amount of water consumed daily during participation in the study, categorized as:
  * 750 mL-1 L
  * 1-1.5 L
  * 1.5-2 L
  * 2 L per day This allows estimation of the participant's hydration level in the 24 hours preceding migraine onset.
Alcohol and/or Substance Use | Daily throughout the 8-week intervention period
  This dichotomous quantitative variable records whether the participant consumed alcohol or other substances within the 24 hours prior to the migraine episode (Yes/No). When "Yes," the type and quantity consumed will be specified
Physical Activity Prior to Migraine Onset | Daily throughout the 8-week intervention period
  This ordinal qualitative variable records whether the participant engaged in physical activity within the 24 hours preceding migraine onset. When physical activity is present, participants may optionally provide a brief description, including perceived intensity and activity type, to help contextualize the potential relationship with migraine triggers.
Moderate/Intense Occupational Activity | Daily throughout the 8-week intervention period
  This nominal quantitative variable records whether the participant performed light, moderate, or vigorous work-related activity during the 24 hours prior to migraine onset, classified according to the World Health Organization (WHO) guidelines on physical activity intensity levels

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad from Sevilla, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study involves personal health information collected under strict confidentiality according to the General Data Protection Regulation (EU) and the Spanish Data Protection Law (LOPDGDD). Only aggregated and anonymized results will be published in scientific journals and repositories.